CLINICAL TRIAL: NCT03800966
Title: A Leaflet-based Programme for Tobacco Industry Denormalisation - a Brief Randomised Controlled Trial
Brief Title: A Brief Intervention Programme for TID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: coshdrama201819
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Attitudes Towards Tobacco Industry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention leaflets will contain information on the TI's tactics to get young people to smoke.
  Interventions: Other: Leaflet
- Control (Placebo Comparator): The control leaflets will contain information on the tobacco control in Hong Kong.
  Interventions: Other: Leaflet

INTERVENTIONS:
Other: Leaflet — Leaflets for both groups will be printed in colour. Leaflet in each group contains 8 pictures and 8 statement, whose sequences will be scrambled. Primary school students need to do the matching, to ensure they read the statements.

SUMMARY:
The brief RCT will be conducted in the form of a questionnaire survey, with two kinds of leaflets embedded in the same questionnaire. The RCT will be conducted in classrooms by teachers who will be given two kinds of questionnaires (with leaflet embedded) used for intervention and control groups. The questionnaires will be mixed in a way that two adjacent questionnaires are always different. The intervention leaflets will contain information for tobacco industry denormalisation. The control leaflets will contain information for tobacco control policy in Hong Kong. The study aims to test the effect of a leaflet-based intervention on primary school students' attitudes towards tobacco industry.

ELIGIBILITY:
Inclusion Criteria:

* Parents and children should all understand Chinese

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Attitudes towards tobacco industry in children | 1 month
  Children will report their opinions towards 4 statements: 1); Tobacco companies are a trustworthy industry; 2) Tobacco industries use many tactics to resist tobacco control regulations; 3) Tobacco industries do everything they can to get young people to smoke; 4) Tobacco industries cheated the public for commercial gain. All the 4 questions have 5 options from definitely yes to definitely no. The options will be recoded into 0-4 or 4-0, as appropriate, with higher scores indicating more negative attitudes towards the industry. A sum of scores from the 4 questions will be deemed as measurement of attitudes towards tobacco industry in primary school students.

SECONDARY OUTCOMES:
Intention to smoke cigarettes in children | 1 month
  Two questions will be used to assess this outcome: 1) If one of your good friends offers you a cigarette, will you smoke it? 2) Do you think you will smoke cigarettes in the next 12 months? Response options are definitely not /probably not /not sure /probably yes /definitely yes. Those choosing options "definitely not" for all the two questions will be deemed having no intention to smoke cigarettes; other responses will be deemed having intention to smoke cigarettes.
Intention to use e-cigarettes in children | 1 month
  Two questions will be used to assess this outcome: 1) If one of your good friends offers you an e-cigarette, will you use it? 2) Do you think you will use e-cigarettes in the next 12 months? Response options are definitely not /probably not /not sure /probably yes /definitely yes. Those choosing options "definitely not" for all the two questions will be deemed having no intention to use e-cigarettes; other responses will be deemed having intention to use e-cigarettes.
Tobacco control policy support in children | 1 month
  Children will report their opinions towards 2 statements: 1) The Hong Kong government should enact a total ban on e-cigarettes promptly; 2) The Hong Kong government should prohibit the sale of all tobacco products by legislation. All the 2 questions have 5 options from definitely yes to definitely no. The options will be recoded into 4-0, with higher scores indicating stronger support towards the tobacco control policy in Hong Kong. A sum of scores from the 2 questions will be deemed as measurement of support for tobacco control policy in Hong Kong in primary school students.
Attitude towards smoking in children | 1 month
  Children will report their opinions towards one statement: Smoking is personal choice, there is no right and wrong. The question has 5 options from definitely yes to definitely no. The options will be recoded into 4-0, with higher scores indicating more negative attitudes towards smoking. Score from that question will be deemed as measurement of attitude towards smoking in primary school students.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided